CLINICAL TRIAL: NCT06936436
Title: the Effect of Implanon on Menstrual Patterns According to Timing of Insertion After Delivery
Brief Title: the Effect of Implanon on Menstrual Patterns
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kholoud Khalid Kamal, OBSTETRICS AND GYNECOLOGY RESIDENT, Assiut University
Other Study IDs: effect of implanon
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Menstrual Irregularities
MeSH Terms: conditions — Menstruation Disturbances | interventions — etonogestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Implanon (Etonogestrel) — implanon is a long acting ,reversible contraceptive implants used to prevent pregnancy

SUMMARY:
This study aims to evaluate whether the timing of postpartum Implanon insertion (immediately postpartum, early postpartum, or late postpartum) affects menstrual patterns

DETAILED DESCRIPTION:
* Etonogestrel implants (Implanon) are widely used for postpartum contraception. However, the timing of insertion may influence menstrual patterns, including irregular bleeding, amenorrhea, and prolonged bleeding episodes. Despite the increasing use of immediate postpartum contraception, there is limited research on how the timing of Implanon insertion affects menstrual cycle regulation.
* Furthermore, lactation and hormonal changes postpartum may modify the bleeding patterns in women using Implanon, with breastfeeding women experiencing a higher likelihood of amenorrhea due to prolactin-induced suppression of ovulation.
* This study aims to fill these gaps by systematically comparing menstrual outcomes based on timing of Implanon insertion postpartum

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women opting for Implanon as contraception.
* No contraindications to hormonal contraception.

Exclusion Criteria:

* . Women with known bleeding disorders.
* Use of other hormonal contraceptives during the study period.
* Postpartum complications such as severe infections or retained products of conception

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Women will be grouped into:
  1. Immediate postpartum (Insertion within 48 hours of delivery).
  2. Early postpartum (Insertion between 4-6 weeks postpartum).
  3. Late postpartum (Insertion after 6 weeks postpartum
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The Effect of Implanon on Menstrual Patterns According to Timing of Insertion After Delivery | baseline
  To compare the effect of Implanon insertion at different postpartum intervals (immediate, early, late) on menstrual cycle patterns
  * To assess the prevalence of irregular bleeding, amenorrhea, and prolonged bleeding across different insertion groups.
  * To analyze general trends in menstrual changes, regardless of insertion timing.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED MOHAMED ABBAS, PROF.DR, Study Chair — Assiut University; MOHAMED SAYED ABDELLAH, PROF.DR, Study Chair — Assiut University; ALAA AHMED MAKHLOUF, DR, Study Chair — Assiut University

REFERENCES:
- [Background] Mazza D, Harrison C, Taft A, Brijnath B, Britt H, Hobbs M, Stewart K, Hussainy S. Current contraceptive management in Australian general practice: an analysis of BEACH data. Med J Aust. 2012 Jul 16;197(2):110-4. doi: 10.5694/mja11.11599. PMID 22794058
- [Background] Richters J, Grulich AE, de Visser RO, Smith AM, Rissel CE. Sex in Australia: contraceptive practices among a representative sample of women. Aust N Z J Public Health. 2003;27(2):210-6. doi: 10.1111/j.1467-842x.2003.tb00810.x. PMID 14696713
- [Background] . Product information: Implanon NXT, Schering-Plough Pty Ltd, 12 November 2010
- [Background] Product information: Implanon® Implant, Organon (Australia) Pty Ltd, 19 March 2008.